CLINICAL TRIAL: NCT05330741
Title: Whole-Body Vibration Versus Gravity Force Stimulation on Postural Stability in Children With Down Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Eman Wagdy, lecturer, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003598
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Down Syndrome
Keywords: Whole-Body Vibration; Gravity Force Stimulation; Biodex Balance System; Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: Designed Physical Therapy program, Whole Body Vibration and, Gravity Force Stimulation
Who Masked: Participant, Outcomes Assessor
Masking Description: By random generator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Designed Physical Therapy Program (Experimental): Designed Physical Therapy Program Down syndrome children will receive the designed physical therapy program for 1 hour. The duration of treatment will be 3 times/week for 12 weeks.
  Interventions: Other: Designed Physical Therapy Program
- Whole-Body Vibration (Experimental): Designed physical therapy program in addition to whole-body vibration. Down syndrome children will receive the designed physical therapy program for 1 hour in addition to whole-body vibration with an amplitude of 2 mm, vibration frequency ranged from 25 to 30 Hz and, vibration time ranged from 5 to10 minutes. The duration of treatment will be 3 times/week for 12 weeks.
  Interventions: Other: Designed Physical Therapy Program; Other: Whole-Body Vibration
- Gravity Force Stimulation (Experimental): Designed physical therapy program in addition to gravity force stimulation. Down syndrome children will receive the designed physical therapy program for 1 hour in addition to gravity force stimulation with 10 repetitions for each position. The duration of treatment will be 3 times/week for 12 weeks.
  Interventions: Other: Designed Physical Therapy Program; Other: Gravity Force Stimulation

INTERVENTIONS:
Other: Designed Physical Therapy Program — The designed physical therapy program include gentle stretching exercises, static muscle contraction, facilitation of trunk control from different positions, balance training from different positions on tilting board, facilitation of righting, protective and equilibrium reactions from different positions, facilitation of standing from different positions, gait training and, climbing stairs up and down.
Other: Whole-Body Vibration — The designed physical therapy program (mentioned before)
  + Whole-body vibration (WBV) training, child will be asked to stand with slightly flexed knees (30 degrees of knee flexion), and both feet will be placed at an equal distance from the center of the platform to achieve an equal distribution of body weight over both feet. The device will set to produce a peak-to-peak sinusoidal vibration with an amplitude of 2 mm and a vibration frequency ranged from 25 to 30 Hz. WBV will applied for (30 sec. of WBV, 1 min rest, 10 repetitions), (45 sec. of WBV, 1 min rest, 10 repetitions), (60 sec. of WBV, 1 min rest, 10 repetitions) in the 1st, 2nd. and 3rd. months respectively.
  Arms: Whole-Body Vibration
Other: Gravity Force Stimulation — The designed physical therapy program (mentioned before)
  + Gravity force stimulation child will be asked to maintain his balance on GFS during each of the following positions as a progression (standing and walking on the surface of two beams connecting the two boxes - standing and walking crossly on the surface of one beam connecting the two boxes - standing and walking sideward on the surface of one beam connecting the two boxes - standing and walking on the edge of the two beams - standing and walking on the edge of one beam: most difficult)
  Arms: Gravity Force Stimulation

SUMMARY:
The purpose of the study is to compare the effect between of whole-body vibration and gravity force stimulation on postural stability in children with Down syndrome.

DETAILED DESCRIPTION:
Down Syndrome (DS) is one of genetic disorders characterized by some common clinical and functional features. Most children with Down syndrome have deficits in postural stability or balance, co-ordination, gait, and functional mobility throughout childhood and adulthood. Postural control dysfunctions are the most common problems found in children with DS leads them to be more inactive, which contributes to functional mobility problems. Several techniques that involve proprioceptive, vestibular, and visual inputs are so beneficial to children with DS. Whole-body vibration (WBV) is one of the training methods that use high-frequency mechanical stimuli generated by a vibrating platform and transmitted through the body, leading to bone loading and sensory receptor stimulation. Gravity force stimulation (GFS) has a strong impact on the child's sensory system helping to normalize the system through exercises that send strong messages to the brain to regulate the tactile, proprioceptive and vestibular components. Hence, there is need to compare between the effects of whole-body vibration training and gravity force stimulation on postural stability in children with Down syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages will be ranged from 8 to 10 years old.
2. Functional hearing and vision.
3. Mild and moderate mental retardation with IQ level (50-70) determined by a psychiatric specialist in the school (IQ measured by Stanford-Binet intelligence scale)
4. Independent standing and walking.

Exclusion Criteria:

1. Synptomatic pain.
2. Musculoskeletal problems or/ atlanto-axial instability.
3. Rheumatic and congenital heart disease
4. History of previous surgical operation
5. Regular participation in any sport activities.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-04-09 (Estimated); Primary Completion 2022-07-09 (Estimated); Study Completion 2022-07-09 (Estimated)

PRIMARY OUTCOMES:
Postural Stability | Up to 12 weeks
  Biodex Stability System will be used to measure overall stability index, anteroposterior stability index and mediolateral stability index.

SECONDARY OUTCOMES:
Functional Mobility | Up to 12 weeks
  Six-minute walk test will be used for measuring functional mobility. It is a sub-maximal test of aerobic capacity, in which the subjects walk as far as possible in 6 minutes (min.) around a premeasured distance